CLINICAL TRIAL: NCT06307756
Title: The Effect of Music Played to Mothers of Premature Babies Inpatient Neonatal Intensive Care Unit on Their Stress Levels and Milk Amount
Brief Title: The Effect of Music on Maternal Stress and Milk Amount
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adiyaman University (Other)
Responsible Party: Principal Investigator, Maksude YILDIRIM, Research Assistant, Adiyaman University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: SayıNo:521
Record Dates: First submitted 2024-02-13; First posted 2024-03-13 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Amount of Breast Milk; Maternal Anxiety Level

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music group (Experimental): Mothers will be informed about the application before the procedure. Mothers who agree to participate in the study will be asked to listen to music that relaxes them for 20 minutes a day for 4 days. The mothers' state anxiety levels and milk quantities will be evaluated before starting the application and every day during the application. Mothers' anxiety levels will be evaluated with the "State Anxiety Inventory". Mothers' anxiety levels and milk quantities will be evaluated every day at 11.45 when they come to the NICU to express milk.
  Interventions: Other: Music group
- Control group (No Intervention): After mothers are informed about the study, mothers who agree to participate in the study will be included in the control group by randomization method. No intervention will be made to mothers in the control group. The mothers' state anxiety levels and milk quantities will be evaluated at the first meeting with the mothers and every day for four days. Mothers' anxiety levels will be evaluated with the "State Anxiety Inventory". Mothers' anxiety levels and milk quantities will be evaluated every day at 11.45 when they come to the NICU to express milk.

INTERVENTIONS:
Other: Music group — Mothers will be informed about the application before the procedure. Mothers who agree to participate in the study will be asked to listen to music that relaxes them for 20 minutes a day for 4 days. The mothers' state anxiety levels and milk quantities will be evaluated before starting the application and every day during the application. Mothers' anxiety levels will be evaluated with the "State Anxiety Inventory". Mothers' anxiety levels and milk quantities will be evaluated every day at 11.45 when they come to the NICU to express milk.
  Arms: Music group

SUMMARY:
Premature babies who have to deal with life-threatening situations have to spend the first days of their lives in intensive care units. Mothers who plan to return home with their babies during the postpartum period may experience stress due to their children being monitored in intensive care. It is stated that mothers of babies in the neonatal intensive care unit experience stress and anxiety due to reasons such as being separated from their babies, the baby's illness, the baby's sensitive body structure, the baby's appearance and behavior, and the baby's dependence on devices. This stress experienced by mothers of premature babies can prevent mothers from providing enough milk to feed their babies. Mothers whose babies are in the neonatal intensive care unit cannot have adequate contact with their babies and cannot breastfeed; It causes insomnia, stress and anxiety, and the hormonal axis is disrupted, negatively affecting the amount of breast milk. In order to support the healing process of preterm babies, it is important to increase the amount of milk produced by mothers and increase the rate at which babies can receive breast milk. Music improves endothelial function by dilating the vessels; It has been reported that it reduces mental stress by increasing the release of nitrite oxide and endorphins and causes many physiological reactions such as a decrease in blood pressure and pulse. This study will examine the effect of music played to mothers with premature babies on maternal anxiety and the amount of breast milk.

ELIGIBILITY:
Inclusion Criteria:

* Mothers whose babies are born prematurely (gestational age between 32-37 weeks), -whose babies do not have any congenital anomalies,
* whose babies are not connected to mechanical ventilation,
* who are over 18 years of age, who are not diagnosed with any psychological disease and
* who agree to participate in the study will be included in the study.

Exclusion Criteria:

* Greater than 32-37 weeks of gestation

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2023-11-15 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-04-22 (Actual)

PRIMARY OUTCOMES:
amount of breast milk measured at the same time every day | 4 months

SECONDARY OUTCOMES:
State Anxiety Inventory | 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- Sağlık Bilimleri Üniversitesi Gazi Yaşargil Eğitim ve Araştırma Hastanesi, Diyarbakır, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No